CLINICAL TRIAL: NCT03455205
Title: The Efficacy and Safety of Shenqi Fuzheng Injection for the Treatment of Cancer-related Fatigue in Chemo Patients With Digestive Tract Were Prospectively, Randomized Blind, Multicenter Clinical Trials
Brief Title: Shenqi Fuzheng Injection for the Treatment of Cancer-related Fatigue in Chemo Patients With Digestive Tract .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Collaborators: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: livzon-sqfz-chemo
Record Dates: First submitted 2017-12-26; First posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2017-12

CONDITIONS: Digestive Tract
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- shenqifuzheng injection (Experimental): Shenqifuzheng injection of 500 ml,intravenous drip, 1 times a day, 7 days post, rest is 14 days, 21 days each for a period of treatment, observation of two procedures. At the same time, according to the NCCN guide and the health ministry issued the diagnosis and treatment guidelines for cancer treatment,The programme provides for chemotherapy regimens:
  Colorectal cancer: CapeOX scheme - oxaliplatin + capecitabine Esophageal cancer: DP/TP programme - docetaxel/paclitaxel + cisplatin/carboplatin Gastric cancer: SOX scheme - oxaliplatin + tigio All test drugs should be covered with dark bags before infusion, and use a dark infusion to guarantee the implementation of the blind method.
  Interventions: Drug: shenqifuzheng
- 0.9% sodium chloride injection (Placebo Comparator): 0.9% sodium chloride injection of 500 ml,intravenous drip, 1 times a day, 7 days post, rest is 14 days, 21 days each for a period of treatment, observation of two procedures. At the same time, according to the NCCN guide and the health ministry issued the diagnosis and treatment guidelines for cancer treatment,The programme provides for chemotherapy regimens: Colorectal cancer: CapeOX scheme - oxaliplatin + capecitabine Esophageal cancer: DP/TP programme - docetaxel/paclitaxel + cisplatin/carboplatin Gastric cancer: SOX scheme - oxaliplatin + tigio No interventions have been included in Arm Description for '0.9% sodium chloride injection'
  Interventions: Drug: 0.9%sodium chloride

INTERVENTIONS:
Drug: shenqifuzheng — 500ml shenqifuzheng daily（at day 1-7and day22-28）through intravenous infusion.
  Arms: shenqifuzheng injection
Drug: 0.9%sodium chloride — 500ml sodium chloride（0.9%）daily（at day 1-7 and day22-28）through intravenous infusion.
  Arms: 0.9% sodium chloride injection

SUMMARY:
The efficacy and safety of cancer patients in patients with gastrointestinal cancer (chemotherapy) in patients with gastrointestinal tumor (chemotherapy) were prospectively, randomized blind, multicenter clinical trials. They were randomly divided into 2 groups, test group Shenqifuzheng injection of 500 ml, the control group 0.9% sodium chloride injection, 500 ml, intravenous drip, 1 times a day, 7 days post, rest is 14 days, 21 days each for a period of treatment, observation of two procedures. At the same time, according to the NCCN guide and the health ministry issued the diagnosis and treatment guidelines for cancer treatment. The main curative effect of the clinic was to evaluate the pretreatment of cancer due to the fatigue score of the patients before and after treatment -- the Piper fatigue revision scale was used to evaluate the Chinese version. Assess effectiveness and safety based on clinical assessment

DETAILED DESCRIPTION:
Factors for the purpose of this study by observing theShenqifuzheng injection before and after treatment in patients with carcinoma due to fatigue scale scores, the classification of syndromes, the quality of life score changes and related laboratory index, evaluation factors ginseng and astragalus injection on the digestive tract tumor (chemotherapy) in patients with cancer-related fatigue and quality of life improved efficacy and safety. The experimental group was randomly divided into 2 groups, experimental group Shenqifuzheng injection of 500 ml. The control group was 0.9% sodium chloride injection, 500ml, intravenous drip, 1 time daily, 7 days for continuous use, 14 days of rest, and 1 treatment for each 21 days, and 2 courses were observed. At the same time, according to the NCCN guide and the health ministry issued the diagnosis and treatment guidelines for cancer treatment.

Main efficacy evaluation indexes before and after treatment for cancer-related fatigue rating - adopting the Piper fatigue scale revised Chinese version, compare the experimental group and the control group before and after treatment cancer-related fatigue rating difference have differences. Secondary efficacy evaluation index to compare the ECOG score difference before and after the treatment, the quality of life score difference before and after the treatment, TCM syndrome curative effect, single symptom curative effect of immune function, tumors had curative effect (if any) and chemotherapy completion. Safety assessment includes the observation of vital signs, blood routine, urinary routine, routine stool, liver function, renal function, electrocardiogram examination, and adverse reactions during the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with gastric cancer, esophageal cancer or colorectal cancer diagnosed by pathology or cytology;
* 2.Diagnostic criteria for cancer-related fatigue;
* 3. Syndrome differentiation of Chinese medicine is a syndrome of lung temper;
* 4. Estimated survival over 3 months;
* 5. ECOG score is less than or equal to 2;
* 6. Age 18 ~ 75 years old;
* 7. Non-surgical indications or reluctance to operate the surgical treatment;
* 8. Have chemotherapeutic indications;
* 9. Stop and chemotherapy for more than 1 month;
* 10. The patient is willing to accept the treatment of the programme, and can follow the doctor's advice to take the medicine and comply with the patient.

Exclusion Criteria:

* 1. The chemotherapy regimen received by the subject was not within the prescribed programme;
* 2. Any situation that may hinder the subject from completing the clinical trial, including but not limited to serious, uncontrollable organic lesions or infection:

  1. clinically significant cardiovascular diseases, such as heart failure (NYHA III-IV), uncontrolled coronary heart disease, cardiomyopathy, arrhythmia, etc.
  2. uncontrolled hypertension (systolic pressure is greater than 160 mmHg or diastolic pressure is greater than 100 mmHg, despite the best drug treatment);
  3. serious clinical infection of activity (greater than 3 degrees NCI-CTCAE 4.03)
  4. severe liver and kidney function abnormality (blood creatinine is greater than 1.5 times ULN; ALT or AST is greater than 2.5 times ULN; Bilirubin is greater than 1.5 times ULN.
* 3. Patients with symptoms, uncontrollable nerves, mental illness or mental disorders;
* 4. Compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2017-12-24 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Piper Fatigue Scale（PFS） | 42 days
  the score of Piper Fatigue Scale before and after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: lin lizhu, Dr., Principal Investigator — First affiliated hospital of guangzhou university of traditional Chinese medicine
Locations (1):
- First affiliated hospital of guangzhou university of traditional Chinese medicine, Guangzhou, Guangdong, China